CLINICAL TRIAL: NCT04524741
Title: Use of Intracardiac Echocardiography or Left Atrial Appendage Radiography to Guide Implantation of a Left Atrial Appendage Occlusion Device.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XieruiqinICE
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Left Atrial Appendage Occlusion

STUDY DESIGN:
Intervention Model Description: A total of 40 patients with atrial fibrillation were scheduled to receive left atrial appendage occlusion, which were divided into two groups. The operation was performed under the guidance of intracardiac echocardiography and left atrial appendage radiography, respectively (allocation ratio 1:1).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- left atrial appendage radiography (Experimental)
  Interventions: Device: intracardiac echocardiography
- intracardiac echocardiography guidance (Experimental)
  Interventions: Device: intracardiac echocardiography

INTERVENTIONS:
Device: intracardiac echocardiography — 30 patients use intracardiac echocardiography to guide left atrial appendage occluder device, 30 patients use radiography to guide left atrial appendage occluder device.
  Other Names: left atrial appendage radiography

SUMMARY:
A total of 40 patients with atrial fibrillation were scheduled to receive left atrial appendage occlusion, which were divided into two groups. The operation was performed under the guidance of intracardiac echocardiography and left atrial appendage radiography, respectively (allocation ratio 1:1). During the operation, the total amount of contrast medium injected, the fluoroscopy time and the time from femoral vein puncture to transseptal puncture to closure were recorded in all patients. The diameter and depth of the left atrial appendage opening were measured by angiography in group A(ICE group), and measured by ICE in group B(radiography group). The size of the occluder device was selected according to the measurement size of the two groups, the occluder device success rate of the two groups was compared, and the relationship between measurement size and the size of the occluder device was obtained.

ELIGIBILITY:
Inclusion Criteria:

patients taking class I and class III antiarrhythmic drugs could not prevent atrial fibrillation, patients younger than 80 years old Cha2ds2-vasc score ≥2 and Has-bled score ≥3, not suitable for long-term oral anticoagulant drugs.

Exclusion Criteria:

Patients with a history of atrial thrombosis or valvular heart disease (moderate or severe valve stenosis or severe valve regurgitation), patients undergoing prosthetic heart valve replacement, pregnant women, patients with previous liver and kidney diseases, malignant tumors or blood system diseases.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
record contrast media as well as fluoroscopy time were recorded | in the procedure
  record contrast media as well as fluoroscopy time were recorded in all patients
measure left atrial appendage opening and depth in different angles by intracardiac echocardiography | in the procedure
  use intracardiac echocardiography to measure left atrial appendage opening and
measure left atrial appendage opening and depth in different angles by radiography | in the procedure
  use left atrial appendage radiography to measure left atrial appendage opening and depth

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China